CLINICAL TRIAL: NCT07069491
Title: Study of Contributing Factors of Intradialytic Hypertension In Hemodialysis Patients at Sohag University Hospitals
Brief Title: Search About Contributing Factors That Leading to Intradialytic Hypertension in Hemodialysis Patients
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aya Ali Amin, Sohag University, Sohag University
Other Study IDs: Soh-Med--25-6-3MS
Record Dates: First submitted 2025-07-04; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Intradialytic Hypertension in Hemodialysis Patients
MeSH Terms: interventions — Sphygmomanometers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Sphygmomanometer — Blood pressure measurement by Sphygmomanometer

SUMMARY:
The aim of this study is searching about contributing factors that leading to intradialytic hypertension in hemodialysis patients more than 18 years old in hemodialysis unit at sohag University hospitals

DETAILED DESCRIPTION:
Study of Contributing Factors of Intradialytic Hypertension in Hemodialysis patients aged more than 18 years old on regular dialysis session for more than 3 months, receiving dialysis session 3 time weekly for 4 hours,blood pressure monitoring for everyone pre and in and post the sessions and records also investigations will be taken before hemodialysis sessions and full medical history will be collected

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 year or older, on maintenance hemodialysis for at least three consecutive, receiving 3 sessions weekly, 4 hours in each session

Exclusion Criteria:

* patients aged less than 18 years old Patients on recent hemodialysis less than 3 months Patients with malignancy, severe infection or sepsis Patients with major bleeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-28 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Study the contributing factors of intradialytic hypertension in hemodialysis patients | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Aya Ali Amin, Study Chair — Sohag University hospitals
Locations (1):
- Faculty of medicine sohag University, sohag Recruiting, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided